CLINICAL TRIAL: NCT04441281
Title: Usability, Safety and Efficacy of AspivixTM, an Atraumatic Innovative Uterine Cervical Traction Device: a Pilot Phase Followed by a Comparative Study (Comparative)
Brief Title: Usability, Safety and Efficacy of AspivixTM (Comparative Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aspivix SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Aspivix_IUD2019_Comparative
Record Dates: First submitted 2020-06-15; First posted 2020-06-22 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: IUD Insertion

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single-blinded - Participants will be blinded towards the intervention used. Additionally, the type of device used will only be revealed to the practitioner after randomization, immediately prior IUD insertion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single-tooth tenaculum (Pozzi forceps) (Active Comparator): In the control arm, a single-tooth tenaculum, Pozzi forceps, used during routine IUD insertion, is employed to hold and stabilize the cervix.
  Interventions: Procedure: Traction of the cervix for IUD insertion
- AspivixTM cervical vacuum tenaculum (Experimental): In the experimental arm, the investigational AspivixTM cervical vacuum tenaculum is employed to hold and stabilize the cervix.
  Interventions: Procedure: Traction of the cervix for IUD insertion

INTERVENTIONS:
Procedure: Traction of the cervix for IUD insertion — Limited mobility of the uterine cervix and alignment with the vaginal canal is often required during insertion of an intrauterine contraceptive device (IUD).

SUMMARY:
Limited mobility of the uterine cervix and alignment with the vaginal canal is often required during insertion of an intrauterine contraceptive device (IUD). Currently, the available instruments are traumatic tenacula, which could cause pain and bleeding and therefore represent an obstacle for certain patients to pursue their medical follow-up.

AspivixTM is a new device, which enables atraumatic traction of the cervix while respecting its specific semi-circular anatomic shape through a system powered by a vacuum chamber.

The aim of our comparative study is to assess the patient's pain and bleeding using the AspivixTM device in comparison with a commonly used single-tooth tenaculum (Pozzi forceps). Additionally, the comparative study aims to assess and compare the safety of the AspivixTM device with the single-tooth tenaculum (Pozzi forceps).

Note: Study is made of 2 phases (pilot phase followed by a comparative phase). Details regarding pilot study is registered separately.

ELIGIBILITY:
Inclusion Criteria:

* Participants older than 18 years
* Participants presenting at the outpatient clinic IUD insertion of Mirena (BAYER), Kyleena (BAYER), Jaydess (BAYER), NOVAT 380 (BAYER), NT Cu380 mini (MONALISA), NT Cu380 (MONALISA), CuT 380A (MONALISA) or CuT 380A QL (MONALISA).
* Participants able to provide informed consent as documented by signature with at least 24 hours of reflection time
* Good understanding of written and oral speaking used at the centre where the study will be carried out.

Exclusion Criteria:

* Participants who are contraindicated for the insertion of the IUD Mirena (BAYER), Kyleena (BAYER), Jaydess (BAYER), NOVAT 380 (BAYER), NT Cu380 mini (MONALISA), NT Cu380 (MONALISA), CuT 380A (MONALISA) or CuT 380A QL (MONALISA).
* Participants under use of excessive alcohol, narcotics or benzodiazepines prior to procedure
* Participants who do not wish to be informed of a chance discovery
* Participant receiving anaesthetics prior to IUD insertion procedure
* Participants on anticoagulant medication
* Participants under use of an analgesic (< 12 hours)
* Previous cervical operation
* Severe vaginal bleeding of unknown origin
* Participant previously enrolled in this study
* Cervix diameter smaller than 26 mm
* Nabothian cyst
* Cervical myomas
* Cervical condylomas
* Squamous intraepithelial lesion (Cervical dysplasia)
* Cervical endometriosis
* Cervical tears
* A well exposed cervix and / or well aligned vaginal and cervical canals where no traction is required for IUD insertion
* Other cervical abnormalities (cervical polyp, cervical lesion, or irregularity) which may contraindicate or complicate IUD insertion
* Large ectopy, for which it is not possible to find a suitable location near the ectopy where native tissue is present
* Large scar tissue, for which it is not possible to find a suitable location near the scar where native tissue is present

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Patient-reported pain: Visual Analogic Scale | Before the procedure
  Patient-reported pain scores (VAS) at specific time points during IUD insertion procedure Minimal and maximal values range from 0 to 100, the higher being the better outcome.
Patient-reported pain: Visual Analogic Scale | During speculum insertion
  Patient-reported pain scores (VAS) at specific time points during IUD insertion procedure Minimal and maximal values range from 0 to 100, the higher being the better outcome.
Patient-reported pain: Visual Analogic Scale | During AspivixTM / standard tenaculum application
  Patient-reported pain scores (VAS) at specific time points during IUD insertion procedure Minimal and maximal values range from 0 to 100, the higher being the better outcome.
Patient-reported pain: Visual Analogic Scale | During application of cervical traction
  Patient-reported pain scores (VAS) at specific time points during IUD insertion procedure Minimal and maximal values range from 0 to 100, the higher being the better outcome.
Patient-reported pain: Visual Analogic Scale | During IUD insertion
  Patient-reported pain scores (VAS) at specific time points during IUD insertion procedure Minimal and maximal values range from 0 to 100, the higher being the better outcome.
Patient-reported pain: Visual Analogic Scale | During AspivixTM / standard tenaculum release
  Patient-reported pain scores (VAS) at specific time points during IUD insertion procedure Minimal and maximal values range from 0 to 100, the higher being the better outcome.
Patient-reported pain: Visual Analogic Scale | 5 minutes after the end of the procedure
  Patient-reported pain scores (VAS) at specific time points during IUD insertion procedure Minimal and maximal values range from 0 to 100, the higher being the better outcome.

SECONDARY OUTCOMES:
The number of placement attempts before traction can be applied | During the procedure to insert the IUD which should last less than 5 minutes.
  number of placement attempts before traction can be applied The number of placement attempts before traction of the cervix can be applied will be recorded
The number of spontaneous releases | During the procedure to insert the IUD which should last less than 5 minutes.
  The number of spontaneous releases during traction of the cervix will be recorded
Assessment of the efficacy of the investigational device and its comparator by the practitioner | During the procedure to insert the IUD which should last less than 5 minutes.
  5 point Likert 'Efficacy Questionnaire' will be used. Minimal to maximal values range from 1 to 5, 1 meaning "disagree" and 5 "agree".
Assessment of bleeding | During the procedure to insert the IUD which should last less than 5 minutes.
  To assess bleeding, every buffer will be weighted, and the blank weight subtracted. Weight in mg will be reported in the case report form.
Assessment of adverse events | During the procedure to insert the IUD which should last less than 5 minutes.
  Safety of the procedure will be assessed by documenting adverse events (description of the adverse events, number of participants)
Assessment of device deficiencies | During the procedure to insert the IUD which should last less than 5 minutes.
  Safety of the procedure will be assessed by documenting device deficiencies (description)
Identification of new risks | During the procedure to insert the IUD which should last less than 5 minutes.
  Safety of the procedure will be assessed by identifying and documenting any new risk.

CONTACTS AND LOCATIONS:
Overall Officials: Patrice Mathevet, Prof., Principal Investigator — DFME CHUV Lausanne
Locations (2):
- Switzerland (2):
  - HUG - Department Women, Child & Adolescent, Geneva, Canton of Vaud
  - Department Women, Mother & Child, University Hospital, Lausanne, Canton of Vaud